CLINICAL TRIAL: NCT07304050
Title: Pilot Randomized Controlled Trial of PICTURE-Pediatric
Brief Title: Randomized Controlled Trial of Predicting Intensive Care Transfers and Other UnfoReseen Events (PICTURE)-Pediatric
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Rodney Daniels, Clinical Associate Professor, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00274862
Record Dates: First submitted 2025-12-23; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Clinical Deterioration
Keywords: Artificial Intelligence model; Usability; Acceptability; Questionnaire; Real-time alerts; Workflow compliance
MeSH Terms: conditions — Clinical Deterioration

STUDY DESIGN:
Intervention Model Description: This study will not be randomization at the patient level. This randomized clinical trial (RCT) will use an on-off design, alternating sequentially between the treatment and control arms on the entire study population. In this design, the model scores and alerts will be available to the care teams for 4 weeks (treatment arm), then the scores will not be available for the following 4 weeks, on for another 4 weeks and so on. Randomization of the first period will be used to minimize bias.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- PICTURE-Pediatric scores and alerts (Experimental): This arm will happen for two four-week periods.
  Interventions: Device: PICTURE-Pediatric scores and alerts
- Control Arm (Other): During the control arm, the PICTURE scores and alerts will not be shown. This arm will happen for two four-week periods.
  Interventions: Other: Control Arm - Scores and alerts hidden

INTERVENTIONS:
Device: PICTURE-Pediatric scores and alerts — Patients that satisfy the inclusion criteria will receive PICTURE-Pediatric scores and alerts. Scores are numbers that indicate the likelihood that the patient may experience deterioration in the next 24 hours, i.e., the higher the score, the higher the likelihood of deterioration. Alerts will be sent through pages or phone notifications, depending on the user's current method of receiving non-routine communications. Scores are also available through electronic medical record as a column that can be wrenched into the patient lists, in a patient summary report and as a vital and/or a flowsheet. The scores for patients with an alert (scores that have surpassed the corresponding alert thresholds) will be colored accordingly (yellow or red) in the electronic medical record. Various staff on the clinical team will use this data to help determine intervention and or escalation depending on the alerts.
  Arms: PICTURE-Pediatric scores and alerts
Other: Control Arm - Scores and alerts hidden — The morning rounds and prerounding procedures will revert back to the baseline procedures before the trial. All care teams will be notified about this transition in advance and will be directed to revert back to the standard of care.
  Arms: Control Arm

SUMMARY:
The purpose of this study is to evaluate the effectiveness and user satisfaction of the study teams early warning system, called PICTURE, which utilizes artificial intelligence (AI) techniques and algorithms to identify patient deterioration on pediatric units within Mott Children's Hospital.

In this pilot study the patient care team will review the PICTURE information and alerts. Morning rounds will be partially informed by the PICTURE scores and the scores will be included in the hand off notes for the patients with a red score.

The primary purpose of this study is to test the hypothesis that the combination of the PICTURE-Pediatric model, the proposed workflow and the proposed interface results in at least 80% compliance.

No participants will be consented as the Institutional review board has approved a waiver of consent for THE clinicians and the patients information being reviewed.

The enrollment numbers will include only the clinicians.

DETAILED DESCRIPTION:
PICTURE Pediatric evaluates large amounts of patient data, labs, monitored data, and vital signs (all variables that are measured as part of routine clinical care and that are stored in the electronic health record in real-time); it does this every 15-minutes and delivers a deterioration risk index score that has been shown to outperform Pediatric Early Warning Score (PEWS), and other similar scoring systems in identifying patients at risk for clinical deterioration. Clinical implementation of PICTURE Pediatric could identify patients at high risk of deterioration early enough to intervene and decrease the need for transfer to the Pediatric Intensive Care unit (PICU), and it could also reduce morbidity and hospital length of stay. This in turn could also improve bed availability for patients awaiting admission in the emergency department and improve efficient transfer out of the PICU, all of which improves care and reduces cost for the patients, their families, and the hospital system.

This protocol also does not mandate or require clinical decisions based on alerts generated (e.g. there is no mandate to transfer to the Intensive Care unit, perform an intervention, or change therapy/clinical course based on PICTURE alerts); rather, the clinical team will decide whether additional investigation, therapy, intervention, or transfer is required after alerts are generated based on staff's clinical experience, knowledge and with consultation with an attending physician when applicable. In case of device failure, there would be no deterioration risk scores generated and the clinical teams would simply continue to follow the current workflow.

ELIGIBILITY:
Inclusion Criteria - Patients:

* Age ≥30 days and ≤25 years
* Be on the general care wards of Mott Children's Hospital or boarding in the Emergency Department (ED), but admitted to a pediatric floor medical team. These will be enforced by these criteria:

  1. Patient class: not emergency b. Patient level of care: not Intensive Care unit (ICU) c. Patient locations (per protocol)

     Exclusion Criteria - Patients:
* Patients that do not meet the inclusion criteria

Ages: 30 Days to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 375 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Compliance with the model workflow as measured by a pop-up questionnaire after each model alert aggregated as a proportion -clinicians | within 30 minutes after each alert during a patient's admission
  Responses to the questions measure compliance with the workflow. Compliance will be measured as binary outcomes (i.e., compliant and noncompliant) and aggregated as a proportion.

SECONDARY OUTCOMES:
Acceptability of Intervention Measure (AIM)-clinicians | At the end of the study (approximately 4 months after the start of the enrollment)
  There are 4 questions that the clinicians will answer about intervention with options from completely agree (5) to completely disagree (1). The range of scores are 4-20 with a higher score indicating greater acceptability.
Intervention Appropriateness Measure (IAM)-clinicians | At the end of the study (approximately 4 months after the start of the enrollment)
  There are 4 questions that the clinicians will answer about intervention with options from completely agree (5) to completely disagree (1). The range of scores are 4-20 with a higher score indicating greater appropriateness.
Feasibility of Intervention Measure (FIM)-clinicians | At the end of the study (approximately 4 months after the start of the enrollment)
  There are 4 questions that the clinicians will answer about intervention with options from completely agree (5) to completely disagree (1). The range of scores are 4-20 with a higher score indicating greater feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Daniels, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No